CLINICAL TRIAL: NCT01196754
Title: Pharmacokinetic of Sevoflurane During a 48h Sedation in ICU With AnaConDa®
Brief Title: Pharmacokinetic of Sevoflurane During a 48h Sedation in Intensive Care Unit With AnaConDa®
Acronym: Anaconda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Estaing (Other)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Purpose: Screening
Other Study IDs: CHU-0079
Record Dates: First submitted 2010-07-15; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Sedation
Keywords: Pharmacokinetics; Sevoflurane; Fluorides; Sedation; Adult patients with a predicted sedation more than 48 h; Stable respiratory and hemodynamic conditions for SBT; Consent of patients; Arterial line
MeSH Terms: interventions — Sevoflurane

ARMS (1):
- sevoflurane (Other)
  Interventions: Other: sevoflurane

INTERVENTIONS:
Other: sevoflurane

SUMMARY:
This is a prospective clinical monocentric study in ICU with sedated ventilated patients with sevoflurane during 48 h with the AnaConda® system, establishing pharmacokinetic model of sevoflurane.

DETAILED DESCRIPTION:
Prospective clinical monocentric study in ICU with sedated ventilated patients with sevoflurane during 48 h with the AnaConda® system, establishing pharmacokinetic model of sévoflurane and its metabolites (hydroxyfluroisopropanol, fluoride)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ventilated more than 48 h
* Stable respiratory and hemodynamic conditions
* Consent of patients or family
* Arterial line

Exclusion Criteria:

* Acute kidney injury
* Obesity
* Sevoflurane anaphylaxia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Determination of plasmatic concentrations of sévoflurane at different times of a 48h sedation of sévoflurane. | during 48 hours

SECONDARY OUTCOMES:
Determination of plasmatic concentrations of HFIP and fluoride at different times of a 48h sedation of sévoflurane. Determination of a pharmacokinetic model of sévoflurane. | during 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bourdeaux, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France